CLINICAL TRIAL: NCT02287441
Title: Feasibility Study Comparing Dietary Methods to Increase Vegetable Consumption
Brief Title: Feasibility Study to Increase Vegetable Consumption
Acronym: VEG1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB2014-090
Record Dates: First submitted 2014-11-06; First posted 2014-11-10 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Increase Intake of Vegetables or Tomatoes; Health
MeSH Terms: interventions — Airway Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raw Group (Placebo Comparator): Vegetables Prepared Raw (raw)
  Interventions: Other: Raw
- Tomato Group (Experimental): Tomato Products (tomato)
  Interventions: Other: Tomato

INTERVENTIONS:
Other: Tomato — Tomato Products (tomato)
  Arms: Tomato Group
Other: Raw — Vegetables Prepared Raw (raw).
  Arms: Raw Group

SUMMARY:
The objective of this study is to determine if differences exist in the total vegetable intake of groups that eat either tomato products versus raw vegetable product.

DETAILED DESCRIPTION:
The proposed study is a crossover 2- arm pilot study comparing vegetable consumption of individuals partaking in two interventions: 1) Tomato Products (tomato) or 2) Vegetables Prepared Raw (raw).

A planned sample size of 20 will be recruited into the study. This study will require one initial screening visit and 5 weekly study visits. This study will take 4 weeks per subject to complete.

The trial will initiate with one screening visit which will last about 1-2 hours where the subjects' height, weight, BMI, waist circumference, fasting glucose, blood pressure and heart rate will be measured along with a survey related to general eating, health and exercise habits.

If willing and eligible to participate, a training of the online 24-hour recall software will be conducted during the screening visit. The subject will then use the software for an upcoming training week to recall foods for 3 days (2 weekdays and 1 weekend).

During the first study visit (End of Week 0) the subject will be randomly assigned an intervention sequence. The intervention sequence will dictate which intervention will be conducted for the first two weeks, leaving the second intervention for the last two weeks. Subjects will receive detailed explanation of their role and types of products they must buy during the upcoming week for the purpose of the study. They will be taught how to record on Vegetable Intake Diaries and be provided with vouchers and coupons to buy study products. They will also be given a recipe book for inspiration during the study to make appropriate meals.

The next study visits (End of Week 1-3) will take place by checking subjects' weight and then providing them with an Experience Questionnaire that is specific to their respective intervention assignment. The questionnaire will ask them to relate their study experiences over the past week. They will return any receipts and labels that were used to buy study products with the vouchers along with completed Vegetable Intake Diary. Before leaving, subjects will be provided with another set of Vegetable Intake Diaries and vouchers.

During Week 2 and 4, subjects will receive 3 surprise notifications (2 weekdays and 1 weekend) to complete the online food records. If they are unable to comply, a different day will be assigned.

The final study visit (End of Week 4) will initiate with anthropometric and vital measurements (height, weight, BMI, heart rate and blood pressure). Subject will complete Experience Questionnaire and return all receipts, labels, and diaries.

The randomization intervention sequence will be randomly assigned based on computer generated sequences. The primary difference between the intervention sequences is the order in which the subject will partake in the two intervention types. While in the tomato intervention, they will be asked to consume extra vegetable through tomato products. While in the raw intervention, however, they can only consume extra vegetables into their diet through raw vegetable products that have not been processed in any way.

Weekly Study Visits will be scheduled approximately 7 days apart.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking men and women ages 25-60 years of age with BMI between 18.5-29.9
* Generally healthy as determined by health history questionnaire
* Weight stable
* Consume a typical western diet
* Access to grocery store with Hunt's tomato products and raw vegetable availability
* Have general cooking skills and kitchen equipped for general food preparation
* Primary shopper and food preparer in household
* Access to internet and ability to complete ASA24
* Past smokers will be allowed in the study if smoking cessation is >1 year (preferred > 2 years).

Exclusion Criteria:

* Smokers
* Current vegetable intake is atypical in type or amount relative to typical American diet
* Currently dieting or taking weight loss medication or weight loss supplements
* Change in weight of more than 5% in the past month
* Special or atypical diet - e.g., vegetarian/vegan, gluten free, excessively high or low energy
* Allergic to common food(s) (dairy, soy, nut/peanut, wheat, intolerance to tomatoes)
* Have fasting blood glucose concentrations >125 mg/dL
* Had cancer other than non-melanoma skin cancer in previous 5 yrs
* Unwilling to eat vegetables
* History of eating disorder or clinical depression as assessed by validated questionnaires.
* Presence of chronic disease or condition (e.g. diabetes, irritable bowel syndrome)
* Chronic or acute gastrointestinal disorder
* Females who are pregnant or breastfeeding
* An athlete in training or highly active person whose dietary intake is greater than average
* Investigator is uncertain about subject's capability or willingness to comply with protocol requirements

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-11-14 (Actual); Primary Completion 2015-05-22 (Actual); Study Completion 2016-04-12 (Actual)

PRIMARY OUTCOMES:
Changes in vegetable and nutrient consumption reported by subject through the 24-Hour online recall software. | 2 weeks
  Changes will be assessed based upon MyPlate.gov serving equivalents for vegetables.

SECONDARY OUTCOMES:
Overall experience with increasing vegetable intake through weekly Experience Questionnaires. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No